CLINICAL TRIAL: NCT01987778
Title: Health Effects of Resistance Training on Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostergotland County Council, Sweden (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Mats Hammar, MD, professor, Ostergotland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20131105/Styrka
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hot Flashes; Menopause
Keywords: Hot flashes; Menopause; HRQoL; Resistance training; Physical activity; Adipose tissue
MeSH Terms: conditions — Hot Flashes; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training (Experimental): The resistance training will be supervised and individualized by an experienced physiotherapist. First the relative load will be lighter during three weeks, thereafter the intensity and load will be increased over another 12 weeks.
  Interventions: Other: Resistance training
- Control group (No Intervention): No intervention for 15 weeks but the same registrations, diaries and forms as the intervention group. The control group will however be omitted from muscle strength testing.

INTERVENTIONS:
Other: Resistance training — Resistance training supervised and individualized by an experienced physiotherapist. First the relative load will be lighter during three weeks, thereafter the intensity and load will be increased over another 12 weeks.
  Arms: Resistance training

SUMMARY:
Today's women will live more than a third of their lives after menopause, i.e. with a changed hormonal and metabolic state. Vasomotor symptoms like hot flushes and sweating are reported by about 75% of all women around menopause and may impair well-being, mental state, daily activities and night sleep. Vasomotor symptoms are less prevalent in women who participate in regular physical exercise. It is, however, still uncertain if physical exercise reduces vasomotor symptoms.

The purpose of this randomized controlled study is to establish possible beneficial health effects from 15 weeks of supervised resistance training (RT) on postmenopausal women. End-points include effects from RT in postmenopausal women on

1. clinical outcomes (number and severity of vasomotor symptoms, Health-Related quality of Life (HRQoL), Body Mass Index (BMI), abdominal height, muscle strength and mass, browning of fat),
2. diagnostic variables (production of myokines as irisin, immunological markers) and
3. genetic variables (length of telomeres).

The control group will be offered resistance training after the intervention period.

DETAILED DESCRIPTION:
The first phase is planned as a pilot-study including 20 women participating for 15 weeks. Thereafter an evaluation of the sample size and the study methodology will be made.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who had at least 28 moderate to severe hot flashes per week during a screening period of two weeks.(Postmenopausal, i.e. had their last menstrual bleeding at least 12 months ago or have increased gonadotrophic hormones showing they are postmenopausal.)
* At lest 45 years of age
* Good physical health and physical ability to take part in organized resistance training or other training at least three times per week.
* Ability to speak and read Swedish
* Freely informed consent for participation

Exclusion Criteria:

* Physically active more than 75 minutes of intense exercise per week or more than 150 minutes of low intensity activities
* Hb <110 g/l
* Blood pressure >160 systolic and/or >100 mmHg diastolic pressure
* Ongoing usage or use during the last two months of hormone therapy aimed for hot flashes
* Treatment with psychopharmacological drugs (e.g SSRI or SNRI) or other treatment with a possible effect on menopausal symptoms
* Uninvestigated or unstable disease that could affect presence of flushes (e.g thyroid disease)
* Other medical condition that is judged inappropriate to combine with physical activity or participation in the study.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in frequency of hot flushes per 24 h | Baseline to 15 weeks of intervention/control group
  Frequency of hot flushes per 24 h daily recorded in hot flush diary from baseline throughout 15 weeks of intervention. Comparison between intervention group and control group.

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL) | Baseline to 15 weeks of intervention/control group. Follow-up after 6 and 24 months.
  HRQoL will be measured with a generic measure (Short Form Health Survey - SF-36) and a measure specifically developed for mid-aged women (Women's Health Questionnaire)
Muscle strength | Baseline to 15 weeks of intervention
  Muscle strength will be evaluated in the intervention group with 8 repetition maximum (8 RM) tests for the major muscles in the extremities.
Level of physical activity | Baseline to 15 weeks of intervention/control group. Follow-up after 6 and 24 months.
  Physical activity will be evaluated using diary and the International Physical Activity Questionnaire (IPAQ).
Concentrations of adipo-myokines/inflammatory biomarkers | Baseline to 15 weeks of intervention/control group
  The markers to assess are as follows: Leptin, Irisin, IL-6, IL-7, IL-8, monocyte chemoattractant protein-1(MCP-1), tumor necrosis factor (TNF), IL-4, IL-10, IL-15, brain-derived neurotrophic factor (BDNF), matrix metalloproteinase (MMP)-2 and MMP-9 in blood samples shortly after a resistance-training and on a day without work-out; samples with direct measurement (plasma) and after white blood cell stimulation, conditioned medium with multiple bead technology (Luminex) and enzyme linked immunosorbent assay (ELISA)
Length of telomeres | Baseline to 15 weeks of intervention/control group
  Length of telomeres will be measured in DNA isolated from blood samples with a qPCR based method. Recently, the telomere length was associated with certain SNP´s in the hTERT gene and these will also be assessed.
Volume of white and brown adipose tissue and muscle volume | Baseline to 15 weeks of intervention/control group
  Using magnetic resonance imaging (MRI) the volume of total (TAT), subcutaneous (SCAT) and visceral (VAT) white adipose tissue (Dahlqvist Leinhard 2008); the concentration of lipids diffusively stored in the liver parenchyma, and the volume of intramuscular adipose tissue (IMAT) in the quadriceps muscle will be quantified. Furthermore, the MRI images will be used to quantify the volume of and fat concentration in supraclavicular and interscapular brown adipose tissue according to our recently published measurement protocol (Lidell 2013, Borga 2013), as well as the volume of the major extensor and flexor muscles (Karlsson 2013).
Body mass index and abdominal height | Baseline to 15 weeks of intervention/control group
  Weight and length (BMI) and abdominal height measured with an abdometer
Blood pressure | Baseline to 15 weeks of intervention/control group
  Using standard measure technique for blood preassure
Severity of hot flushes | Baseline to 15 weeks of intervention/control group. Follow-up after 6 and 24 months.
  Severity of hot flushes per 24 h recorded in hot flush diary from baseline throughout 15 weeks of intervention and one week during follow-up at 6 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mats L Hammar, Professor, Principal Investigator — Linkoeping University
Locations (1):
- County Council of Östergötland, Kvinnokliniken, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahlqvist Leinhard O, Johansson A, Rydell J, Smedby Ö, Nyström F, Lundberg P, Borga M. Quantitative Abdominal Fat Estimation Using MRI. 2008 19th International Conference on Pattern Recognition, ICPR 2008 , art. no. 4761764.
- [Background] Lidell ME, Betz MJ, Dahlqvist Leinhard O, Heglind M, Elander L, Slawik M, Mussack T, Nilsson D, Romu T, Nuutila P, Virtanen KA, Beuschlein F, Persson A, Borga M, Enerback S. Evidence for two types of brown adipose tissue in humans. Nat Med. 2013 May;19(5):631-4. doi: 10.1038/nm.3017. Epub 2013 Apr 21. PMID 23603813
- [Background] Borga M, Virtanen KA, Romu T, Leinhard OD, Persson A, Nuutila P, Enerback S. Brown adipose tissue in humans: detection and functional analysis using PET (positron emission tomography), MRI (magnetic resonance imaging), and DECT (dual energy computed tomography). Methods Enzymol. 2014;537:141-59. doi: 10.1016/B978-0-12-411619-1.00008-2. PMID 24480345
- [Background] Karlsson A, Rosander J, Tallberg J, Romu T, Borga M, Dahlqvist Leinhard O. Whole Body Muscle Classification using Multiple Prototype Voting. Proceedings of the ISMRM Annual Meeting (ISMRM'13), 2013.
- [Background] Daley A, Stokes-Lampard H, Macarthur C. Exercise for vasomotor menopausal symptoms. Cochrane Database Syst Rev. 2011 May 11;(5):CD006108. doi: 10.1002/14651858.CD006108.pub3. PMID 21563149
- [Background] Beavers KM, Brinkley TE, Nicklas BJ. Effect of exercise training on chronic inflammation. Clin Chim Acta. 2010 Jun 3;411(11-12):785-93. doi: 10.1016/j.cca.2010.02.069. Epub 2010 Feb 25. PMID 20188719
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Ivarsson T, Spetz AC, Hammar M. Physical exercise and vasomotor symptoms in postmenopausal women. Maturitas. 1998 Jun 3;29(2):139-46. doi: 10.1016/s0378-5122(98)00004-8. PMID 9651903
- [Background] Kim JH, Ko JH, Lee DC, Lim I, Bang H. Habitual physical exercise has beneficial effects on telomere length in postmenopausal women. Menopause. 2012 Oct;19(10):1109-15. doi: 10.1097/gme.0b013e3182503e97. PMID 22668817
- [Background] Lindh-Astrand L, Nedstrand E, Wyon Y, Hammar M. Vasomotor symptoms and quality of life in previously sedentary postmenopausal women randomised to physical activity or estrogen therapy. Maturitas. 2004 Jun 15;48(2):97-105. doi: 10.1016/S0378-5122(03)00187-7. PMID 15172083
- [Background] Taylor JD, Fletcher JP. Reliability of the 8-repetition maximum test in men and women. J Sci Med Sport. 2012 Jan;15(1):69-73. doi: 10.1016/j.jsams.2011.07.002. Epub 2011 Aug 5. PMID 21820961
- [Derived] Nilsson S, Henriksson M, Hammar M, Berin E, Lawesson SS, Ward LJ, Li W, Holm AS. A 2-year follow-up to a randomized controlled trial on resistance training in postmenopausal women: vasomotor symptoms, quality of life and cardiovascular risk markers. BMC Womens Health. 2024 Sep 13;24(1):511. doi: 10.1186/s12905-024-03351-1. PMID 39272114
- [Derived] Nilsson S, Hammar M, West J, Borga M, Thorell S, Spetz Holm AC. Resistance training decreased abdominal adiposity in postmenopausal women. Maturitas. 2023 Oct;176:107794. doi: 10.1016/j.maturitas.2023.107794. Epub 2023 Jul 6. PMID 37421844
- [Derived] Berin E, Spetz Holm AC, Hammar M, Lindh-Astrand L, Bertero C. Postmenopausal women's experiences of a resistance training intervention against vasomotor symptoms: a qualitative study. BMC Womens Health. 2022 Jul 30;22(1):320. doi: 10.1186/s12905-022-01900-0. PMID 35907840